CLINICAL TRIAL: NCT01679743
Title: A Pilot Study of GRN1005 for Resectable Brain Metastases in Patients With Breast Cancer and Non-Small Cell Lung Cancer
Brief Title: GRN1005 for Brain Metastases From Breast or Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 120199; 12-C-0199
Record Dates: First submitted 2012-09-01; First posted 2012-09-06 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2014-08-11

CONDITIONS: Breast Cancer; Lung Neoplasms; Breast Neoplasms; Lung Cancer
Keywords: Metastatic Breast Cancer; Metastatic Lung Cancer; Monoclonal Antibody; 18FLT; Surgery
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Trastuzumab

ARMS (2):
- A (Experimental): Breast Cancer Cohort
  Interventions: Drug: Trastuzumab; Drug: GRN 1005
- B (Experimental): Non-Small Cell Lung Cancer Cohort
  Interventions: Drug: GRN 1005

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be administered after GRN1005 in patients with HER2+ metastatic breast cancer.
  Arms: A
Drug: GRN 1005 — GRN1005 will be administered at a dose of 550 mg/m2 as an IV infusion at a rate of 8.0 - 8.5 mL/minute on Day 1 of 21-day cycle ( 3 days) and a second dose will be given on the day of surgery (day 21) 3-6 h prior to surgery.

SUMMARY:
Background:

- Brain metastases are cancer cells that have spread to the brain from primary cancers in other organs. These tumors can be removed surgically. However, researchers are trying to find better ways to treat brain metastases. A new drug, GRN1005, has been designed to cross into the brain and deliver the cancer treatment drug paclitaxel to treat tumors. Researchers want to see how well GRN1005 works on brain metastases from breast or lung cancer.

Objectives:

- To test the safety and effectiveness of GRN1005 in treating brain metastases from breast or lung cancer.

Eligibility:

- Individuals at least 18 years of age who have breast or lung cancer that has spread to the brain.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Tumor tissue samples may also be collected. Imaging studies will also be performed.
* Participants who have breast cancer will be divided into two groups. Those whose cancer contains the HER2 protein will be treated with the drug Herceptin as well as GRN1005. Those without HER2 will have only GRN1005.
* Participants who have lung cancer will also have only GRN1005.
* All participants will have two doses of GRN1005, each 3 weeks apart. On the day the second dose of GRN1005 is given, participants will undergo surgery to remove the brain tumors.
* Treatment will be monitored with frequent blood tests and imaging studies.

DETAILED DESCRIPTION:
Background:

Brain metastasis is the most common intra-cranial tumor in adults with approximately 170,000 new cases being diagnosed in the United States annually. The incidence of brain metastasis is increasing. Usually brain metastases of breast cancer occur after the diagnosis of systemic metastases; but approximately 10 25% of patients with lung cancer have brain metastases at diagnosis and another 40 50% develop them during the course of their disease. Multiple factors are contributing to this increase: aging population, improved imaging techniques, and improvement in the treatment of tumors leading to prolonged survival, thereby allowing the emergence of brain metastases, with the brain being generally regarded as a sanctuary site because of the blood brain barrier (BBB). Lung cancer and breast cancer are the leading tumor types, accounting for approximately 50% and 15 - 20% of patients with brain metastases. This study will evaluate the ability of 18F-FLT to determine if amount of change in the uptake in the brain metastases from breast and lung cancer after one dose of therapy with GRN1005, correlates with intra-cranial response. FLT-PET utilizes a radiolabeled form of thymidine, which is incorporated into DNA in proliferating cells. 18F-FLT uptake correlates better than 18F-FDG with proliferation, tumor progression, and survival. Because CNS uptake of FLT is low in contrast to FDG, this makes it potentially useful in evaluating CNS metastases. We would like to see which of these imaging modalities is superior in detection of brain metastases, and monitoring response to therapy.

Objectives:

-Determine whether one cycle of therapy GRN1005 is associated with a change in FLTPET uptake.

Eligibility:

* Adult patients (greater than or equal to 18 years)
* Histologically or cytologically-documented breast cancer (HER2 status must be known) or NSCLC
* Presence of resectable brain metastases based on evaluation by neurosurgery.
* At least one radiologically-confirmed and measurable metastatic brain lesion.

Design:

* Pilot non-randomized trial with or without trastuzumab
* Ten patients with resectable brain metastases from breast cancer and ten patients with resectable brain metastases from NSCLC will be studied.
* Baseline imaging (brain tumor protocol MRI and DSC-PWI MRI, FLT-PET) 1-14 days prior to first dose of GRN1005.
* Patients will receive 1 dose of GRN1005 on day 1 of study.
* Repeat FLT-PET imaging and MRIs will be done after 1 cycle of therapy and prior to surgery, on day 21.
* On the day of surgery, patients will receive a second dose of GRN1005 3 to 6 hours prior to brain surgery.
* PK studies will be done after each dose of GRN1005.
* Optional extra-cranial tumor biopsies will be performed before and after GRN1005 administration.
* Following surgery radiation therapy will be offered to patients as clinically indicated per radiation oncologist s recommendation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult patients (greater than or equal to 18 years)
* Histologically or cytologically-documented breast cancer (HER2 status must be known) or NSCLC
* Presence of resectable brain metastases with or without prior radiotherapy. Patients must be greater than 28 days from WBRT or SRS
* Presence of resectable brain metastases, as assessed by neurosurgical evaluation. A brain tumor will be considered to be resectable for the purposes of the study if it is located in the cerebrum or the cerebellum. Tumors that are located in deep brain structures, including the medulla, pons, midbrain, thalamus, and basal ganglia will be considered non-resectable. The tumor must be solitary or, if not, accompanied by another tumor on the same side of the brain that is also considered to be resectable by the same criteria.
* At least one radiologically-confirmed and measurable metastatic brain lesion (greater than or equal to 1.0 centimeters in the longest diameter) by Gd-MRI of the brain less than 14 days prior to first dose of GRN1005 (Cycle 1, Day 1). The spatial resolution of the Philips Gemini TOF PET/CT is 4millimeters [FWHM, (full width half maximum)]. One cm is greater than 2 times this FWHM and it is anticipated that greater than 70% of the actual activity in the lesion will be visualized (i.e. recovered). It is expected that all lesions greater than or equal to 1 centimeters will have sufficient FLT uptake. If no lesions on the baseline image are visualized on FLT PET/CT, then post therapy FLT imaging will not be performed. These patients will be replaced.
* Patients must be neurologically stable, defined as being on stable doses of corticosteroids and anticonvulsants (not enzyme-inducing antiepileptic drugs (EIAEDs), including phenytoin, phenobarbitol, carbamazepine, fosphenytoin, primidone, oxcarbazepine) for greater than or equal to 5 days prior to obtaining the baseline Gd-MRI of the brain and greater than or equal to 5 days prior to first dose of GRN1005
* Karnofsky Performance Score (KPS) greater than or equal to 80% (which is equivalent to Eastern Cooperative Oncology Group [ECOG] Performance Status of 0 or 1)
* Life expectancy greater than 3 months
* Completed cytotoxic chemotherapy greater than or equal to 21 days (for an every 3-week regimen) or greater than or equal to 14 days (for an every 2-week or weekly regimen) prior to first dose of GRN1005 (Cycle 1, Day 1); all clinically significant toxicities (excluding alopecia) must have resolved to less than or equal to CTCAE v4.0 Grade 1.
* Completed treatment with non-cytotoxic systemic drugs (e.g., targeted drugs) greater than or equal to 14 days for small molecules and greater than or equal to 28 days for monoclonal antibodies (e.g., bevacizumab, with the exception of trastuzumab and bisphosphonates) prior to first dose of GRN1005 (Cycle 1, Day 1). All clinically significant toxicities (excluding alopecia) must have resolved to less than or equal to CTCAE v4.0 Grade 1.
* Adequate laboratory test results for organ systems less than equal 14 days prior to first dose of GRN1005, as follows:

  * Absolute neutrophil count (ANC) greater than or equal to 1.5 times 10(9)/L
  * Hgb greater than or equal to 9.0 grams per deciliter
  * Platelets greater than or equal to 100 times 10(9)/L
  * Total bilirubin less than 1.6 milligrams per deciliter or less than the upper limit of normal (ULN). Serum bilirubin less than 2 times ULN for patients with Gilbert s syndrome
  * Aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT;

SGPT) less than 2.5 times ULN. AST, ALT less than 5 times ULN for patients with documented liver metastases

* Alkaline phosphatase less than 2.5 times ULN. For patients with documented liver or bone metastases, alkaline phosphatase less than 5 times ULN
* Serum creatinine less than 1.5 milligrams per deciliter or creatinine clearance greater than or equal to 45 millliter per minute

  * Negative pregnancy test less than or equal to 72 hours prior to Cycle 1, Day 1 of GRN1005 (for all women of reproductive potential)
  * Patients with HER2-positive disease who are on trastuzumab should be willing and able to continue receiving trastuzumab in accordance with standard institutional practice and prescribing information (EF greater than or equal to 50 % and no history of trastuzumab related CHF or greater than or equal 16% absolute decrease in LVEF from pre-treatment values or an LVEF value below institutional limits of normal and greater than or equal 10% absolute decrease in LVEF from pretreatment values). If these criteria are not met, trastuzumab will not be administered during this protocol.
  * Ability of subject or Legally Authorized Representative (LAR) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study.

EXCLUSION CRITERIA:

* NCI CTCAE v4.0 Grade greater than or equal to 2 neuropathy
* CNS disease requiring immediate neurosurgical intervention (e.g., resection, shunt placement, etc.)
* Known leptomeningeal disease
* Known severe hypersensitivity or allergy to paclitaxel or any of its components
* Treatment with P450 CYP 3A4 or 2C8 enzyme-inducing anticonvulsant drugs less than or equal to 14 days prior to first dose of GRN1005 (Cycle 1, Day 1)
* Patients with the presence of an infection including abscess or fistulae, or infection with hepatitis B or C or HIV
* Any evidence of severe or uncontrolled systemic disease, such as clinically significant cardiovascular (including arrhythmias), pulmonary, hepatic, renal, or metabolic disease; wound-healing disorders; ulcers; or bone fractures
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of clinically significant interstitial lung disease on chest CT scan
* Severe conduction disturbance including clinically significant QTc prolongation defined as a QTc greater than 450 milliseconds in women and QTc greater than 440 milliseconds in men (unless pacemaker in place).
* Women or men of reproductive potential not consenting to use double-barrier contraceptive methods (e.g., diaphragm plus condom) or abstinence during the study, from screening until 3 months after the last GRN1005 administration, and if applicable, for 6 months after the last trastuzumab administration
* Women who are pregnant or breast-feeding
* Prior GRN1005 treatment
* Allergy to gadolinium used in MRI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08-29; Primary Completion 2014-08-11 (Estimated); Study Completion 2014-08-11 (Estimated)

PRIMARY OUTCOMES:
Effect of GRN therapy on PET uptake after treatment cycle 1 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Platta CS, Khuntia D, Mehta MP, Suh JH. Current treatment strategies for brain metastasis and complications from therapeutic techniques: a review of current literature. Am J Clin Oncol. 2010 Aug;33(4):398-407. doi: 10.1097/COC.0b013e318194f744. PMID 19675447
- [Background] Steeg PS, Camphausen KA, Smith QR. Brain metastases as preventive and therapeutic targets. Nat Rev Cancer. 2011 May;11(5):352-63. doi: 10.1038/nrc3053. Epub 2011 Apr 7. PMID 21472002
- [Background] Lagerwaard FJ, Levendag PC, Nowak PJ, Eijkenboom WM, Hanssens PE, Schmitz PI. Identification of prognostic factors in patients with brain metastases: a review of 1292 patients. Int J Radiat Oncol Biol Phys. 1999 Mar 1;43(4):795-803. doi: 10.1016/s0360-3016(98)00442-8. PMID 10098435